CLINICAL TRIAL: NCT00100204
Title: Salivary Proteomics in Disease and Health
Brief Title: Salivary Proteins in Disease and Health
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050058; 05-D-0058
Record Dates: First submitted 2004-12-23; First posted 2004-12-24 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-04-19

CONDITIONS: Diabetes Mellitus; Sarcoidosis; Dental Caries; Sjorgren's Syndrome; Cystinosis; Head and Neck Neoplasms
Keywords: Head and Neck Radiation; Diabetes; Sarcoidosis; Sjogren's Syndrome; Caries; Healthy Volunteer; HV; Saliva Sample
MeSH Terms: conditions — Diabetes Mellitus; Sarcoidosis; Dental Caries; Cystinosis; Head and Neck Neoplasms; Sjogren's Syndrome

SUMMARY:
This study will examine saliva samples from healthy volunteers and patients with various diseases to learn more about how disease affects the mouth and salivary glands. It will use a method called salivary proteomics to identify multiple proteins in saliva and discover if there are protein patterns unique to specific diseases. The study will:

* Characterize the salivary proteome in patients with Sjogren's syndrome, graft-versus-host disease, diabetes, sarcoidosis, cystinosis, dental caries, and immunodeficiencies and in patients who have had head and neck radiation
* Evaluate the possible use of salivary proteomics for early diagnosis
* Evaluate the potential use of salivary proteomics for prognosis and treatment

Patients participating in NIH clinical studies who have Sjogren's syndrome, graft-versus-host disease, diabetes, sarcoidosis, cystinosis, dental caries, or an immunodeficiency, or patients undergoing head and neck radiation may be eligible for this study. Candidates are screened with a medical and dental history, head and neck examination, and photographs of any mouth sores or disease. Healthy volunteers also have blood drawn for routine laboratory testing.

Participants have saliva collected from the floor of the mouth, the parotid salivary glands in the cheek, and the submandibular and sublingual salivary glands under the tongue. Patients with certain diseases also provide a urine sample. Saliva samples are collected as follows:

* One time from healthy volunteers and patients with Sjogren's syndrome, diabetes, sarcoidosis, cystinosis and immunodeficiencies
* Five times from patients undergoing stem cell transplant: at baseline before transplant and about 1, 2, 3 and 6 months after transplant.
* Three times from patients undergoing head and neck radiation: at baseline before radiation and at 3 and 6 months after the conclusion of radiation.

DETAILED DESCRIPTION:
The diagnostic potential of the proteomic methods has been explored by several groups in recent years. Saliva contains many proteins, some of which are altered in various disease states. In this study, saliva is to be sampled in patients with head and neck radiation, diabetes, hematopoietic stem cell transplant, Sjogren's syndrome, cystinuria, methylmalonic acidemia and other conditions. Various novel analytical and data-processing tools will be used to infer characteristic salivary protein and salivary analyte signatures of these disorders. In some cases, these data will be evaluated with data for the oral flora present in the saliva and plaque of these patient groups and relate the presence and levels of particular bacteria to the proteomic profile.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Male and female subjects of all ages and racial groups will be included. The lower age limit will be determined by the ability to cooperate with saliva collection methods: i.e. 6 months to 100 years old.
  2. Patients will be recruited from current NIH Clinical Center pools or the outside community. Patients must be diagnosed with cystinosis, sarcoidosis, head and neck cancer, Sjogren's syndrome or diabetes by their institute physician. Controls will be recruited from various NIH populations who are generally healthy and without one of the diseases listed above or through the NIH Healthy Volunteer Program.
  3. Patients with both benign and malignant disease undergoing bone marrow transplant or hematopoeitic stem cell transplant will be eligible. Among patients with malignant disease both solid tumors and leukemias will be included. Patients who can be diagnosed unequivocally with GVHD via biopsy of the affected organ system will be included in the disease group. Patients will be included in control group when GVHD can be reliably excluded.
  4. For caries studies, we will examine salivary samples already collected from a large twin cohort study in Brazil. These samples were collected from twins and their siblings as part of a study of early childhood caries. Results from that study suggest that genetics has a role in the development of caries. Whole salivary samples have been collected and frozen for further analysis. These samples will be examined for differences in salivary proteins which may be associated with the development of early childhood caries. Samples are coded with a unique numerical identifier with clinical diagnosis for caries, as well as subject age, gender and ethnicity. No other patient information is linked to this identifier to ensure patient confidentiality.

EXCLUSION CRITERIA:

1. Patients receiving autologous HCT or peripheral stem cell transplants.
2. Patients unable to cooperate with saliva collection.
3. Controls with a medical history or laboratory findings consistent with Sjogren's syndrome, sarcoidosis, diabetes, or generally poor health, or controls taking medications known to alter salivary protein profiles.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2004-12-21; Study Completion 2011-04-19

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Fusaro VA, Stone JH. Mass spectrometry-based proteomics and analyses of serum: a primer for the clinical investigator. Clin Exp Rheumatol. 2003 Nov-Dec;21(6 Suppl 32):S3-14. PMID 14740422
- [Background] Hanash S. Disease proteomics. Nature. 2003 Mar 13;422(6928):226-32. doi: 10.1038/nature01514. PMID 12634796
- [Background] Pusch W, Flocco MT, Leung SM, Thiele H, Kostrzewa M. Mass spectrometry-based clinical proteomics. Pharmacogenomics. 2003 Jul;4(4):463-76. doi: 10.1517/phgs.4.4.463.22753. PMID 12831324